CLINICAL TRIAL: NCT05123274
Title: Mobilizing Social Network Resources for HIV Care Support: Development and Testing of an Intervention for HIV+ MSM in St. Petersburg, Russia
Brief Title: Mobilizing Social Network Resources for HIV Care Support
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Yuri A. Amirkhanian, PhD, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH125715 (NIH)
Record Dates: First submitted 2021-11-04; First posted 2021-11-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Care Counseling (Active Comparator): After completing the baseline survey, each participant will receive a 20-minute individual counseling session focused on HIV medical care. The session will convey that effective HIV treatment is now available at no cost, protects health, and that most individuals who are in treatment can lead long and healthy lives. Referral will be made and assistance provided in accessing LGBT-friendly HIV medical care, mental health, substance abuse, and other services.
  Interventions: Behavioral: Individual Care Counseling
- Social Support Mobilization (Experimental): In addition to the post-baseline 20-minute individual counseling session, each participant in this arm will attend five main intervention sessions and two booster sessions that have three inter-related objectives: (1) ensuring that participants understand that viral suppression through ART maintains health and protects others; (2) increasing resilience and feelings of self-worth; and (3) guiding participants in identifying, accessing, and mobilizing social resources for both general psychosocial support and also specific supports for HIV care. For individuals who have potential supports in their social environment, the intervention will seek to mobilize or increase the frequency and quality of interactions with them. For participants who are presently socially isolated or whose social resources are not supportive of HIV care, the intervention will help to build new social ties with potentially supportive life figures.
  Interventions: Behavioral: Social Support Mobilization

INTERVENTIONS:
Behavioral: Social Support Mobilization — Five main sessions and two booster sessions focused on providing accurate information about HIV medical care, increasing participants' feelings of resilience and self-worth, and mobilizing or creating social supports.
  Other Names: SSM
  Arms: Social Support Mobilization
Behavioral: Individual Care Counseling — Twenty-minute individual counseling session focused on HIV medical care
  Arms: Individual Care Counseling

SUMMARY:
The intervention study will recruit 100 out-of-care HIV+ men who have sex with men in online and in community settings located throughout St. Petersburg, Russia. After completing baseline assessments, participants will be randomized to either an individual care counseling (ICC) comparison condition or ICC plus a social support mobilization (SSM) intervention. In each intervention, participants will attend five main and two booster sessions that underscore the benefits of medical care engagement, counter the effects of internalized intersectional stigma and promote resilience, and help participants develop and mobilize social resources supportive of HIV care. Support mobilization will begin by assisting participants develop care-supportive bonds with other group members, friends who are also living with HIV, and connections made with LGBT and other non-governmental organizations. They will also be guided in developing and expanding supportive links with affirmative friends, family members, and other resources. In this way, the intervention will bolster care-related social support resources, resilience, and feelings of self-worth. Assessments administered at baseline will be repeated 6 and 12 months post-intervention, and in-depth followup interviews will be conducted with a subset of 20 participants to elicit feedback about the intervention experience. The study will investigate whether the SSM intervention will produce greater preliminary evidence of benefit on the primary outcome of medical care attendance in the past 6 months and on secondary outcomes of having undetectable viral load, ART adherence, and psychosocial well-being.

DETAILED DESCRIPTION:
100 HIV+ men who have sex with men (MSM) will be recruited and will complete an individual baseline assessment of HIV medical care engagement, adherence if prescribed antiretroviral medications, substance use, psychosocial well-being, social resources, and a blood draw for viral load testing. At the end of the baseline visit, participants will receive counseling about HIV care as well as referral for medical care and other services. The 100 participants will be randomized to one of two conditions. 50 participants will receive only the counseling provided during the baseline visit (ICC Comparison Group). The 50 participants assigned to the experimental condition will additionally receive the Social Support Mobilization (SSM) intervention being tested in the research. A subset of 20 intervention attendees will participate in in-depth followup interviews to elicit their feedback about the intervention experience. All study participants will complete 6- and 12-month followup assessments with measures administered at baseline. If there is evidence of intervention benefit, members of the former comparison condition will be offered the intervention after the final followup point as an ethical service.

Participant Recruitment

St. Petersburg is a large city with a population of 4.5 million residents. Participants will be recruited from:

1. venues such as support groups and events held by non-governmental organizations;
2. virtual spaces such as HIV+ and gay-oriented online forums, boards, and social media sites; and
3. through community announcements in venues where MSM meet.

The use of multiple modalities for recruitment in a large city will result in a sample of HIV+ MSM with minimal potential for overlap. Interested individuals will be asked to contact the study office by telephone or social media. Ineligible persons will be referred for HIV medical and other services. Individuals whose HIV status is not confirmed by baseline testing will be excluded.

Baseline Assessment Procedures and Measures. All study activities will take place at a community-based office located in central St. Petersburg, easily accessible by public transportation. Eligible participants will provide written informed consent at the start of the 90-minute individual baseline assessment session.

Demographic characteristics and health history. Participants will provide information about their demographic characteristics (age, income, education, and relationship status) and HIV-related health history (length of HIV+ serostatus knowledge and HIV care, treatment, and ART history).

HIV care engagement, appointment keeping, and ART adherence. Respondents will be asked how many HIV-related medical treatment appointments they attended in the past 6 months; how many appointments were scheduled, kept, or missed; and date of their most recent appointment. Russian HIV care providers give patients a document that specifies the date of their most recent medical visit and test results. To verify treatment attendance, participants will be asked to bring the document to their assessment visit. For participants prescribed anti-retroviral therapy, two adherence measures will be administered: (1) the Visual Analog Scale (VAS) completed to indicate percentage of medication doses taken as prescribed in the past month, shown valid for measuring adherence; and (2) the HRSA SPNS ART Adherence Scale, a measure with well-established reliability and validity.

HIV viral load testing. A blood sample drawn by the project's physician or nurse will be tested to verify serostatus and determine HIV viral load, considered undetectable if <200 copies/ml., a cutoff based on prior research findings. Viral load testing biologically corroborates care and adherence self-reports.

Measures of medication-taking readiness and self-efficacy. Participants not on anti-retroviral medication therapy will be administered 9 items of the HIV Medication Readiness Scale (sample item: "How ready are you to accept the idea of taking HIV pills for a long time?"). Participants ever prescribed anti-retroviral medication therapy will complete the HIV Medication-Taking Self-Efficacy Scale that consists of two subscales, Self-Efficacy Beliefs (sample item: "How confident are you in your ability to take HIV medication at correct intervals?") and Outcome Expectancies (sample item: "Taking HIV medication will allow you to live a long life").

Scales of psychosocial well-being. To determine if the planned intervention benefits participants' psychosocial adjustment, participants will complete the Social Provisions Scale to measure perceived social supports; the Center for Epidemiological Studies-Depression to measure depression; and the State Anxiety Inventory. Stigma associated with HIV and with same-sex orientation will also be measured. The HIV Stigma Scale assesses overall HIV stigma and personalized stigma, disclosure concerns, negative self-image, and concern with public attitudes. The Homosexuality-Related Stigma Scale measures experienced and internalized stigma associated with same-sex behavior.

Transmission risk behavior and substance use. The level of alcohol use and problem drinking will be assessed by presenting a list of alcohol and illicit drugs commonly used in Russia and asking participants on how many days in the past month each was used and how much was used on the day of greatest use. Participants reporting drug injection will be asked about type of drug, frequency of injection, and use of clean needles. Participants will report on their number and types of male and female sex partners in the past 3 months, frequency of condomless intercourse, and HIV concordance by partner.

Assessment of social resources. Levels and change over time in participants' number and quality of supportive relationships will be measured using the Social Network Map originally developed and validated, and shown to have strong psychometric characteristics by Tracy and Whittaker. Content will be adapted to also assess HIV care support. Respondents list, by first name and last name initial, individuals in their lives who provide emotional support, practical assistance, financial assistance, socializing and advice/guidance. The Social Network Map yields a total network size score as well as scores for network size in each of the domain-specific areas. Use of this instrument will determine whether the intervention produces change in number of social resources over time and in the perceived quality of support from them.

Individual care-related counseling session. After completing all measures, each participant will receive a 20-minute individual counseling session focused on HIV medical care conducted by project staff who hold master's degrees in counseling-related fields carefully trained to protocol.

Sessions will always convey that effective HIV treatment is now available at no cost, protects health, and that most people living with HIV and in treatment can lead long and healthy lives. Referral will be made and assistance provided in accessing LGBT-friendly HIV medical care, mental health, substance abuse, and other services.

Randomization of Participants to Study Conditions. Following baseline data collection, the participants will be randomly allocated in equal numbers by the study biostatistician to one of the two study conditions.

Intervention Procedures.

Individual care counseling (ICC)-only comparison condition. All study participants will receive the baseline individual counseling session described above. This constitutes the only intervention provided to comparison condition participants.

Social Support Mobilization (SSM) Intervention. The study's intervention is based on the hypothesis that participants who have social supports will obtain better outcomes. Thus, the intervention will teach and guide participants in identifying, accessing, and mobilizing social supports.

Intervention Conduct. Groups of 8 to 10 participants will attend five weekly sessions followed by booster sessions to sustain momentum two and again four weeks after the main intervention. Each session will last for about 2-1/2 hours and be led by an experienced 2-member team of facilitators who hold Master's degrees in behavioral/social sciences and are experienced in facilitating HIV-related group sessions with MSM. Staff who conduct intervention sessions will always be different than those who recruit, consent, and assess participants. Groups will be close-ended and scheduled at a time convenient for all members. The same group of participants will attend the full series of intervention sessions together in order to build mutual supports and cohesion. Individuals who miss a session will be offered the opportunity to attend a make-up session.

The intervention has three inter-related objectives: (1) ensuring that participants understand that viral suppression through ART maintains health and protects others; (2) increasing resilience and feelings of self-worth; and (3) guiding participants in identifying, accessing, and mobilizing social resources for both general psychosocial support and also specific supports for HIV care. For individuals who have potential supports in their social environment, the intervention will seek to mobilize or increase the frequency and quality of interactions with them. For MSM who are presently socially isolated or whose social resources are not supportive of HIV care, the intervention will help to build new social ties with potentially supportive life figures.

The intervention will assist participants in mobilizing mutual supports for HIV care with other session participants, with other HIV+ friends, and through involvement in the programs, activities, and message boards of LGBT and community advocacy organizations in St. Petersburg. Bonds formed through these channels are likely to be accepting, affirmative, and nonjudgmental. Participants will discuss, practice, and plan ways to offer-and ways to gain-care-related informational supports (such as sharing information about care providers known to be affirmative and accessible), emotional supports (helping one another cope with life stressors), and tangible supports (helping one another get to clinic appointments). Intervention sessions will link group members to mutually support one another in care-related strategies, and will assign participants to reach out to other friends or to the programs of LGBT organizations where they can link with others for care supports. Beyond supports specific to HIV care engagement, the intervention will also seek to build social resources for general psychosocial well-being and for social integration with persons believed to be supportive of health and self-esteem.

Sessions will employ interactive discussion, skills-building exercises, group problem solving, and goal-setting for social support mobilization and for mutual care-related supports. Week-by-week, participants will be asked to share with one another challenges and care barriers they face, life concerns they have, steps taken toward HIV care engagement, and social connections made since the last session. In these ways, the intervention will help participants develop and mobilize social capital that can directly support HIV care engagement and also strengthen psychosocial well-being.

All participants who received the SSM intervention will complete measures eliciting intervention feedback at the end of the final booster session. In addition, 40% of participants will be randomly selected for in-depth interviews to provide feedback and discuss their experience in the intervention and perceptions about how it can be improved. The interviews will be conducted immediately after the intervention ends so that participants' memories will be fresh. The interviews will seek feedback on all aspects of the intervention including its most and least useful format, content and interactive techniques, and outcomes of social resource mobilization efforts. Interviews will delve into reactions of others to participants' social resource mobilization efforts. Interviews will be conducted by experienced in-depth interviewers uninvolved in intervention delivery, will be recorded, and will be thematically analyzed.

Followup Assessment Procedures. Participants will be followed at points 6 and 12 months after the final main intervention session with assessments that include all behavioral measures administered at baseline as well as viral load testing. Followups will also measure how often in the past month the participant talked with friends about HIV care topics. These questions will determine whether there were changes over time in care-supportive talk among participants across the study conditions.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* male at birth
* reports being HIV-positive with no HIV medical care visit in the prior 6 months or adhering to <95% of ART medication in the past month
* reports a history of sex with males in the prior 12 months
* not a participant in the earlier pilot test of the intervention

Exclusion Criteria:

* age 17 or younger
* not male at birth
* reports being HIV-negative or unknown HIV status
* reports being HIV-positive with at least one HIV medical care visit in the prior 6 months or reports adherence to >95% of prescribed ART in the past month
* reports no history of sex with males in the prior 12 months
* participation in the earlier pilot test of the intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
HIV Medical Appointments Kept | 6 months
  The number of HIV medical care appointments a participant has attended
HIV Medical Appointments Missed | 6 months
  The number of HIV medical care appointments a participant has missed

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States